CLINICAL TRIAL: NCT02159937
Title: In Vitro Functional Modulation of Monocyte-derived Dendritic Cells of Patients With Cancer by Peptides
Status: Completed | Type: Observational
Sponsor: Recepta Biopharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PDCX
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Cancer
Keywords: cancer; in vitro; peptides; dendritic cells
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with metastatic cancer: Blood sampling by vena punction.
  Interventions: Other: Blood sampling by vena punction.

INTERVENTIONS:
Other: Blood sampling by vena punction. — In vitro tests will be performed after blood sample collection from metastatic cancer patients

SUMMARY:
The purpose of this study is to evaluate in vitro the potential of peptides, to modify, phenotypically and functionally, the monocyte-derived dendritic cells of patients with metastatic cancer.

DETAILED DESCRIPTION:
The DCs will be generated in vitro from peripheral blood mononuclear cells (PBMCs) which will be obtained from 30 ml of peripheral blood collected from each patient with metastatic cancer by venipuncture in heparin tubes.

The cellular viability, the expression of maturation biomarkers and the presence of several cytokines will be evaluated by flow cytometric assays after the culture period of DCs exposed to the peptides.

An interim analysis is programmed with the first 10 patients. If an effect is demonstrated the study will include an additional number of subjects sufficient to ensure adequate comparison with other commercially available peptides.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of the Informed Consent Form before the performing of any procedures related to the study;
2. Age ≥18 years;
3. Histologically confirmed metastatic malignant neoplasia;
4. Results of laboratorial exams in the first 6 weeks before the blood sample collection within the following values:

   * White blood cells ≥ 3.000/μL;
   * Platelet count ≥ 100,000/mm³;
   * Hemoglobin > 10g/dL;
   * Serum aspartate aminotransaminase (AST), alanine aminotransferase (ALT) and alkaline phosphatase < 2.5 x upper limit of normal (ULN);
   * Serum creatinine < 1.5 x upper limit of normal (ULN);
5. Karnofsky performance status ≥ 70%.

Exclusion Criteria:

1. Presence of autoimmune disorders or conditions that require systemic treatment with immunosuppressant medications or systemic corticosteroids;
2. Received any systemic chemotherapy or radiotherapy within 15 days prior to the blood sample collection;
3. Received any immunotherapy within 4 weeks prior to the blood sample collection;
4. Known history of positive serology for HIV (human immunodeficiency virus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed metastatic malignant neoplasia.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Expression of cellular markers in the dendritic cells (DCs) after stimulation with the peptides. | At the seventh day of the cells culture period
Viability of the dendritic cells (DCs) after stimulation with the peptides. | At the seventh day of the cells culture period
Cytokines production by the dendritic cells (DCs) after stimulation with the peptides. | At the seventh day of the cells culture period

CONTACTS AND LOCATIONS:
Overall Officials: José AM Barbuto, Ph.D, Study Chair — Departamento de Imunologia - Instituto de Ciências Biomédicas da Universidade de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil